CLINICAL TRIAL: NCT02605187
Title: Patient-Driven Analgesic Protocol Selection for Post-Cesarean Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brendan Carvalho, Chief, Division of Obstetric Anesthesia Department of Anesthesiology, Perioperative and Pain Medicine, Stanford University School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 34740
Record Dates: First submitted 2015-11-10; First posted 2015-11-16 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Postoperative Pain
Keywords: cesarean; postoperative pain; patient choice
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Acetaminophen; Gabapentin; Morphine; Matrilin Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- No choice (Active Comparator): No choice given medium dose intrathecal morphine acetaminophen po q6h ibuprofen po q6h
  Interventions: Other: No choice given; Drug: Ibuprofen; Drug: Acetaminophen; Drug: Morphine (med)
- Choice: low protocol (Experimental): Choice given low dose intrathecal morphine acetaminophen po q6h ibuprofen po q6h
  Interventions: Other: Choice given; Drug: Ibuprofen; Drug: Acetaminophen; Drug: Morphine (low)
- Choice: medium protocol (Experimental): Choice given medium dose intrathecal morphine acetaminophen po q6h ibuprofen po q6h
  Interventions: Other: Choice given; Drug: Ibuprofen; Drug: Acetaminophen; Drug: Morphine (med)
- Choice: high protocol (Experimental): Choice given high dose intrathecal morphine acetaminophen po q6h ibuprofen po q6h gabapentin po one time dose
  Interventions: Other: Choice given; Drug: Ibuprofen; Drug: Acetaminophen; Drug: Gabapentin; Drug: Morphine (high)

INTERVENTIONS:
Other: No choice given — Patients are randomized to getting a choice or not getting a choice. If they do not get a choice, they receive standard dose.
  Arms: No choice
Other: Choice given — Patients are randomized to getting a choice or not getting a choice. If they do get a choice, they will receive the protocol they select.
  Arms: Choice: high protocol; Choice: low protocol; Choice: medium protocol
Drug: Ibuprofen — Ibuprofen 600mg po q6h
Drug: Acetaminophen — Acetaminophen 650mg po q6h
Drug: Gabapentin — Gabapentin 600mg po one time within 1 hour of delivery
  Arms: Choice: high protocol
Drug: Morphine (low) — Intrathecal morphine dose 50mcg
  Other Names: Low dose morphine
  Arms: Choice: low protocol
Drug: Morphine (med) — Intrathecal morphine dose 150mcg
  Other Names: Medium dose morphine
  Arms: Choice: medium protocol; No choice
Drug: Morphine (high) — Intrathecal morphine 300mcg
  Other Names: High dose morphine
  Arms: Choice: high protocol

SUMMARY:
The ability to predict pain and then apply modified treatment protocols has been limited. Current practice is for physicians to select standard post-operative pain treatment protocols without patient consultation. This study hopes to determine if patient's involvement in analgesic drug/dosage selection can optimize pain relief while minimizing related side effects. This could result in a more patient-centered care model and individualized perioperative analgesic treatment protocols based on patient's preferences, needs and expectations.

DETAILED DESCRIPTION:
This randomized, controlled study will include a simple, preoperative questionnaire to obtain baseline demographic and obstetric data; and complete questions (that have previously been shown to be predictive of postoperative pain) from which we will determine their expected and target postoperative pain scores. These questionnaires should take less than 3-4 minutes to complete.

The subject will then be randomized into "choice" and "no choice" groups. The randomization for choice vs. no choice will be at a 1:3 ratio i.e. 1 woman will get no choice and 3 will get a choice for their analgesic protocol. All women will receive the same medications for intraoperative anesthetic management -- only the postoperative pain medications will be altered.

The no choice group will receive the current standard analgesic protocol: medium dose intrathecal morphine, and around the clock acetaminophen po q6h and ibuprofen po q6h.

The group with the choice will be offered 3 different protocols:

1. low dose intrathecal morphine, and around the clock acetaminophen po q6h and ibuprofen po q6h. 2 medium dose intrathecal morphine, and around the clock acetaminophen po q6h and ibuprofen po q6h. 3. high dose intrathecal morphine, and around the clock acetaminophen po q6h and ibuprofen po q6h, as well as gabapentin po one time within 1 hr of delivery.

Women randomized to the "choice" group will select a protocol after being given a standard script explaining advantages and disadvantages of each protocol.

Drugs and doses utilized in the study are safe for postpartum women and within dose range routinely used at our and other institutions.

All breakthrough pain will be managed the same for all patients, and adequate analgesia will be available to treat post-operative pain.

Primary breakthrough rescue analgesic will be our standard oral opioid oxycodone managed using our current treatment algorithm. If pain 1-4 out of 10, 1 tablet (5 mg) will be offered, if pain >4 out of 10, 2 tablets (10 mg) will be offered PRN. Pain not responding to oral opioids will be offered IV morphine boluses or PCA as per standard treatment protocols. Additional analgesic options (e.g. TAP blocks) will also be available as per standard care.

Following standard Cesarean delivery, postoperative data will be collected (directly from patients and from the electronic medical record) by study investigators blinded to group assignment.

Outcome measures:

1. Pain scores at rest and on to sitting (VPS 0-10) collected at 3, 6, 12, 24, 36, 48 hours post-cesarean
2. Overall daily pain score and its deviation from target and expected pain score will be determined at 0-24 and >24-48 hours study periods.
3. Opioid use (oral and IV morphine) in the 0-24 and >24-48 hour study periods.
4. Time to first analgesic for breakthrough pain (minutes from spinal)
5. Side effect: Pruritus score (0-100), nausea score (0-100) and number of episodes of vomiting for the 0-24 and >24-48 hour post- operative periods
6. Any treatment of pruritus and/or nausea/vomiting
7. Satisfaction with postoperative analgesia score (0-100)
8. Discharge time (hours/minutes from surgery end)

Telephone follow-up for pain score, opioid use, and functional recovery will be performed at 1 week, 1 month, 3 months and 6 months post-Cesarean. The telephonic questions will last 3-4 minutes

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-50
* Singleton gestation
* Not in active labor
* Scheduled for their 1st, 2nd, or 3rd elective Cesarean
* Cesarean deliveries under spinal or combined spinal epidural anesthesia (with no additional epidural doses administered)

Exclusion Criteria:

* History of chronic pain, anxiety, or depression
* Unable to understand the concept of Verbal Numerical Pain Scale at the time of informed consent
* Chronic consumption of opiates, antidepressants or anticonvulsants
* Intake of opioids, NSAIDS or acetaminophen 48hrs prior to the psychophysical test
* Preeclampsia (with any severe features)
* Diabetes (not controlled with diet and needing drugs)
* Preterm delivery (<35 weeks gestation)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, MBBCh, MDCH, Principal Investigator — Stanford University
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

REFERENCES:
- [Background] Eisenach JC, Pan P, Smiley RM, Lavand'homme P, Landau R, Houle TT. Resolution of pain after childbirth. Anesthesiology. 2013 Jan;118(1):143-51. doi: 10.1097/ALN.0b013e318278ccfd. PMID 23249931
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Lavand'homme P. Perioperative pain. Curr Opin Anaesthesiol. 2006 Oct;19(5):556-61. doi: 10.1097/01.aco.0000245284.53152.1f. PMID 16960491
- [Derived] Carvalho B, Sutton CD, Kowalczyk JJ, Flood PD. Impact of patient choice for different postcesarean delivery analgesic protocols on opioid consumption: a randomized prospective clinical trial. Reg Anesth Pain Med. 2019 May;44(5):578-585. doi: 10.1136/rapm-2018-100206. Epub 2019 Mar 13. PMID 30867278

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Started | 40 | 21 | 83 | 16
Completed | 32 | 19 | 72 | 15
Not Completed | 8 | 2 | 11 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol | Total
Number analyzed (Participants) | 32 | 19 | 72 | 15 | 138
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [32 to 39] | 37 [34 to 39] | 34 [32 to 36] | 33 [30 to 36] | 35 [31 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 19 | 72 | 15 | 138
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 19 | 11 | 42 | 11 | 83
  Asian | 9 | 7 | 27 | 3 | 46
  Other | 4 | 1 | 3 | 1 | 9
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 28 [27 to 31] | 28 [25 to 30] | 29 [26 to 33] | 30 [28 to 35] | 28 [26 to 33]
Gestational age (week) [Median (Inter-Quartile Range); unit: week] | 39.0 [39.0 to 39.1] | 39.1 [39.1 to 39.4] | 39.0 [39.0 to 39.4] | 39.0 [39.0 to 39.2] | 39.0 [39.0 to 39.4]
Education [Count of Participants; unit: Participants]
  High school | 4 | 1 | 3 | 2 | 10
  Some college | 5 | 1 | 8 | 2 | 16
  BA or equivalent | 10 | 3 | 28 | 6 | 47
  Graduate Degree | 13 | 14 | 33 | 5 | 65
Nulliparous [Count of Participants; unit: Participants] | 4 | 6 | 16 | 3 | 29
Previous Cesarean Delivery [Count of Participants; unit: Participants] | 21 | 15 | 45 | 10 | 91
Language [Count of Participants; unit: Participants]
  English | 27 | 19 | 66 | 11 | 123
  Other | 5 | 0 | 6 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption in the 0-48 Hour Study Periods.
Description: Opioid consumption was measured in milligram morphine equivalents in the 0-24 and 24-48 hour study periods.
Time Frame: 0-24 and 24-48 hour postoperative periods
Population: Participants who completed the protocol are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: milligram morphine equivalents (MMEQ)
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
milligram morphine equivalents (MMEQ)
  0-24 hours | 10 [0 to 15] | 5 [0 to 20] | 10 [0 to 25] | 5 [0 to 30]
  24-48 hours | 10 [0 to 30] | 0 [0 to 10] | 5 [0 to 20] | 30 [10 to 40]

2. Primary Outcome: Pain Scores
Description: Pain scores at rest and at movement post-cesarean delivery. Score was rated on a scale from 0 to 10, where 0=no pain and 10=worst imaginable pain.
Time Frame: 3, 6, 12, 24, 36 and 48 hours after delivery
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
units on a scale
  Pain at rest at 3 hours | 1.6 (2.0) | 1.8 (2.0) | 1.9 (2.1) | 2.2 (2.2)
  Pain at movement at 3 hours | 3.2 (2.9) | 3.4 (2.5) | 3.2 (2.7) | 4.1 (2.5)
  Pain at rest at 6 hours | 2.3 (2.3) | 2.7 (1.9) | 2.2 (1.8) | 1.5 (1.6)
  Pain at movement at 6 hours | 4.0 (2.7) | 4.4 (2.4) | 3.8 (2.4) | 3.8 (2.4)
  Pain at rest at 12 hours | 1.5 (1.7) | 2.1 (1.7) | 1.9 (1.8) | 1.7 (1.7)
  Pain at movement at 12 hours | 3.0 (2.3) | 4.7 (1.5) | 3.6 (2.0) | 3.2 (2.1)
  Pain at rest at 24 hours | 2.2 (1.9) | 1.9 (1.0) | 2.2 (1.7) | 2.3 (1.7)
  Pain at movement at 24 hours | 4.5 (2.3) | 4.1 (1.5) | 4.3 (2.0) | 3.6 (1.8)
  Pain at rest tat 36 hours | 1.5 (1.6) | 1.7 (1.3) | 2.6 (2.0) | 3.1 (2.4)
  Pain at movement at 36 hours | 3.5 (2.2) | 4.0 (2.1) | 4.5 (2.0) | 4.8 (1.8)
  Pain at rest at 48 hours | 1.7 (1.6) | 2.0 (1.9) | 2.0 (1.6) | 3.3 (2.2)
  Pain at movement at 48 hours | 3.5 (1.9) | 3.9 (1.8) | 3.6 (1.8) | 4.8 (2.5)
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of pain at rest 24 hours after delivery. Null Hypothesis: all the means are the same; Test type: Superiority; p = 0.882, ANOVA — Final parameter estimates would be considered significant at P < 0.05
Statistical Analysis 2: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of pain at movement 24 hours after delivery. Null Hypothesis: all the means are the same; Test type: Superiority; p = 0.565, ANOVA — Final parameter estimates would be considered significant at P < 0.05
Statistical Analysis 3: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of pain at rest 48 hours after delivery. Null Hypothesis: all the means are the same; Test type: Superiority; p = 0.022, ANOVA — Final parameter estimates would be considered significant at P < 0.05
Statistical Analysis 4: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of pain at movement 48 hours after delivery. Null Hypothesis: all the means are the same; Test type: Superiority; p = 0.140, ANOVA — Final parameter estimates would be considered significant at P < 0.05

3. Secondary Outcome: Count of Participants Who Need Opioid Use
Description: Count of participants who need opioid use through 48 hours after delivery.
Time Frame: 0-24 and 24-48 hours after delivery
Population: Participants who completed the protocol are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
Participants
  0-24 hours after delivery | 27 | 14 | 50 | 13
  24-48 hours after delivery | 23 | 8 | 42 | 14
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of opioid use 0-24 hours after delivery; Test type: Superiority; p = 0.311, Fisher Exact — Final parameter estimates would be considered significant at P < 0.05
Statistical Analysis 2: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of opioid use 24-48 hours after delivery; Test type: Superiority; p = 0.008, Fisher Exact — Final parameter estimates would be considered significant at P < 0.05

4. Secondary Outcome: Count of Participants With Presence of Pruritus
Description: Count of participants with pruritus through 48 hours after delivery.
Time Frame: 0-24 and 24-48 hours after delivery
Population: Participants who completed the protocol are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
Participants
  0-24 hours after delivery | 27 | 11 | 63 | 13
  24-48 hours after delivery | 12 | 3 | 29 | 7
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of presence of pruritus 0-24 hours after delivery; Test type: Superiority; p = 0.092, Fisher Exact
Statistical Analysis 2: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of presence of pruritus 24-48 hours after delivery; Test type: Superiority; p = 0.269, Fisher Exact

5. Secondary Outcome: Pruritus Score at 24 and 48 After Delivery
Description: Score was rated on a scale from 0 to 10, where 0=no itching and 10=most itching.
Time Frame: 24 and 48 hours following delivery
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
units on a scale
  24 hours after delivery | 4.2 (2.7) | 1.7 (2.3) | 3.7 (2.5) | 4.5 (2.7)
  48 hours after delivery | 0.8 (1.3) | 0.2 (0.6) | 1.0 (1.8) | 1.1 (1.4)
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of pruritus score 24 hours after delivery. Null Hypothesis: all means are equal; Test type: Superiority; p = 0.006, ANOVA
Statistical Analysis 2: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of pruritus score 48 hours after delivery. Null Hypothesis: all means are equal; Test type: Superiority; p = 0.296, ANOVA

6. Secondary Outcome: Count of Participants Who Need Medical Treatment of Pruritus
Description: Count of participants who need medical treatment of pruritus during first 48 hours after delivery.
Time Frame: 0-24 and 24-48 hours after delivery
Population: Participants who completed the protocol are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
Participants
  0-24 hours after delivery | 7 | 2 | 12 | 3
  24-48 hours after delivery | 2 | 0 | 2 | 0
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of participants who need medical treatment of pruritus 0-24 hours after delivery; Test type: Superiority; p = 0.759, Fisher Exact
Statistical Analysis 2: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of participants who need medical treatment of pruritus 24-48 hours after delivery; Test type: Superiority; p = 0.761, Fisher Exact

7. Secondary Outcome: Counts of Participants With Presence of Nausea
Description: Count of participants with nausea through 48 hours after delivery.
Time Frame: 0-48 hours after delivery
Population: Participants who completed the protocol are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
Participants | 11 | 7 | 33 | 10
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Test type: Superiority; p = 0.281, Chi-squared

8. Secondary Outcome: Nausea Score Score at 24 and 48 After Delivery
Description: Score was rated on a scale from 0 to 10, where 0=no nausea and 10=most nausea.
Time Frame: 0-24 and 24-48 hours after delivery
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
units on a scale
  0-24 hours after delivery | 1.3 (2.4) | 1.1 (2.0) | 1.5 (2.4) | 1.8 (1.7)
  24-48 hours after delivery | 0.3 (0.9) | 0.2 (0.5) | 0.2 (0.7) | 0.2 (0.6)
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of nausea score 24 hours after delivery. Null Hypothesis: all means are equal; Test type: Superiority; p = 0.786, ANOVA
Statistical Analysis 2: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of nausea score at 48 hours after delivery. Null Hypothesis: all means are equal; Test type: Superiority; p = 0.985, ANOVA

9. Secondary Outcome: Counts of Participants Who Need Medical Treatment for Nausea
Description: Counts of participants who need medical treatment of nausea through 48 hours after delivery.
Time Frame: 0-24 and 24-48 hours after delivery
Population: Participants who completed the protocol are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
Participants
  0-24 hours after delivery | 8 | 9 | 20 | 9
  24-48 hours after delivery | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of participants who need nausea treatment from 0-24 hours after delivery; Test type: Superiority; p = 0.057, Chi-squared
Statistical Analysis 2: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of participants who need nausea treatment from 24-48 hours after delivery; Test type: Superiority; p = 0.246, Fisher Exact

10. Secondary Outcome: Average Number of Vomiting Episodes After Delivery
Time Frame: 0-24 and 24-48 hours after delivery
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: vomiting episodes
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
vomiting episodes
  0-24 hours after delivery | 0.6 (1.5) | 0.3 (1.0) | 0.5 (1.4) | 1.3 (2.0)
  24-48 hours after delivery | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of average number of vomiting episodes 0-24 hours after delivery. Null Hypothesis: all means are equal; Test type: Superiority; p = 0.226, ANOVA

11. Secondary Outcome: Time to Discharge
Description: Minutes from delivery until discharge.
Time Frame: Delivery through discharge (average 4 days)
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
minutes | 4771.9 (1231.2) | 4652.1 (1006.7) | 5278.9 (1410.3) | 5722.3 (1391.9)
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Test type: Superiority; p = 0.036, ANOVA

12. Secondary Outcome: Patient Overall Satisfaction With Postoperative Analgesia
Description: Score was rated on a scale from 0 to 100, where 0=completely unsatisfied and 100=completely satisfied.
Time Frame: 24 and 48 hours after delivery
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
Number analyzed (Participants) | 32 | 19 | 72 | 15
units on a scale
  24 hours after delivery | 87.2 (12.7) | 90.3 (10.4) | 94.1 (9.5) | 93.3 (7.7)
  48 hours after delivery | 89.9 (10.6) | 92.6 (9.7) | 91.2 (15.1) | 89.3 (14.0)
Statistical Analysis 1: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of satisfaction with pain medication 24 hours after delivery; Test type: Superiority; p = 0.019, ANOVA
Statistical Analysis 2: Comparison: No Choice vs Choice: Low Protocol vs Choice: Medium Protocol vs Choice: High Protocol; Comparison of satisfaction with pain medication 48 hours after delivery; Test type: Superiority; p = 0.873, ANOVA

ADVERSE EVENTS:
Time Frame: Delivery to discharge (average 4 days)
Arm/Group | No Choice | Choice: Low Protocol | Choice: Medium Protocol | Choice: High Protocol
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/19 | 0/72 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/19 | 0/72 | 0/15
Other Adverse Events (participants affected / at risk) | 3/32 | 1/19 | 6/72 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Choice (N=32) | Choice: Low Protocol (N=19) | Choice: Medium Protocol (N=72) | Choice: High Protocol (N=15)
Pain due to Bakri balloon and vag pack (Surgical and medical procedures) | 1 | 0 | 0 | 0
received methergine for Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 1
Itching rash on abdomen (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Migrain (Nervous system disorders) | 0 | 1 | 0 | 0
Severe pre E diagnosed postpartum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
misoprostol used at delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Vomit (General disorders) | 0 | 0 | 1 | 0
preeclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Surrogate (General disorders) | 0 | 0 | 1 | 0
Urinary Tract Infections (Infections and infestations) | 0 | 0 | 1 | 0
Used On Q pump (General disorders) | 0 | 0 | 0 | 1
Extended stay (General disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT02605187/Prot_SAP_000.pdf